CLINICAL TRIAL: NCT03375229
Title: Dry Needling and Photobiomodulation in the Treatment of Myofascial Pain
Brief Title: Dry Needling and Low-level Laser Therapy to Treat Myofascial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Rafael Inácio Barbosa, Principal Investigator, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1205-4687
Record Dates: First submitted 2017-12-05; First posted 2017-12-18 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Myofascial Pain; Trigger Points
Keywords: Myofascial Pain; Pain Pressure Threshold; Low-Level Laser Therapy; Dry Needling
MeSH Terms: interventions — Dry Needling; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group On (Active Comparator): This group was composed of 15 subjects. The application of dry needling and Low-Level Laser Therapy (LLLT) turned on will be directly on the trigger point. The intervention will be administered one time.
  Interventions: Other: Dry Needling; Device: Low-Level Laser Therapy
- Group Off (Active Comparator): This group was composed of 14 subjects. The application of dry needling and LLLT turned off will be directly on the trigger point. The intervention will be administered one time.
  Interventions: Other: Dry Needling; Device: Low-Level Laser Therapy
- Placebo group (Placebo Comparator): This group was composed of 14 subjects. The application of dry needling and LLLT turned off will be 1.5 cm medially from the trigger point. The intervention will be administered one time.
  Interventions: Other: Dry Needling; Device: Low-Level Laser Therapy

INTERVENTIONS:
Other: Dry Needling — It will be used acupuncture needles, individually packaged and sterilized, with 0.25 mm of thickness and 0.40 mm of length. The therapist will perform the grip in upper trapezius on the site of one of the two previously marked locations, according to the subject group allocation, and will insert the needle in the skin with help of a guide tube and will deepen the needle approximately 10 to 15 mm inside the trigger point. The needle will be moved up and down as in the "fast-in and fast-out" technique described by Hong and the movement will be repeated during 30 seconds in a cadence of approximately 1 Hz. The protocol will be the same for the groups that will receive the application directly on the trigger point and for the group that will receive the application away from the trigger point
Device: Low-Level Laser Therapy — The laser protocol used the PainAway Laser™ cluster equipment composed of one pulsed infrared laser of 905 nm, four red LEDs of 640 nm, and four infrared LEDs of 875 nm, with full device aperture of 4 cm2, total delivered energy of 39,8 J, a magnetic field of 35 Mt and treatment time of 300 seconds. The equipment was turned on only for the DNP group and it remained in slight contact with the skin during 300 s for all groups.
  Other Names: LLLT

SUMMARY:
Myofascial Pain is a clinical condition of myalgic pain characterized mainly by the presence of Myofascial Trigger Points. Trigger points can be active or latent and they are described as a hypersensitive spot within a taut band in the muscle. The use of a computer for long periods has been shown as a trigger the trigger points. Dry Needling and Low-Level Laser Therapy (LLLT) has been described as good resources to treat myofascial pain. The hypothesis is that the association of the purposed interventions will have greater effects than only the dry needling intervention. The objective is to evaluate the effects of the dry needling and the laser in the treatment of upper trapezius trigger point on women. This study is composed of an evaluation and an intervention proposal with dry needling and LLLT to treat myofascial trigger points. The sample will be composed of 60 women, with 18 to 65 years old, divided into three groups. Twenty individuals will be in group Dry-On that will receive dry needling intervention on the trigger point, followed by LLLT intervention on. Twenty individuals will be in group Dry-Off that will receive dry needling intervention on the trigger point, followed by LLLT intervention turned off. Twenty individuals will be in group Control that will receive dry needling intervention at 1.5 cm from the trigger point, followed by LLLT intervention turned off. All interventions will be performed in one session. Outcome measures for pain, pressure pain threshold, functionality, and muscle activity will be collected.

DETAILED DESCRIPTION:
The present study has the objective to evaluate the effects of dry needling and photobiomodulation application in the treatment of trigger points in upper trapezius on women with myofascial pain. The specific objectives are: 1) To evaluate the pain level before, during, and after the dry needling and photobiomodulation applications on the trigger point; 2) To identify the pain pressure threshold before and after dry needling and photobiomodulation applications on the trigger point; 3) To verify the electromyographic activity of upper trapezius before and after the proposed treatments; and 4) To compare the effects fond intra and inter-groups for the applications of dry needling, dry needling and photobiomodulation, and control protocol.

The sample will be composed by 20 subjects in each group, a total of 60 subjects, according to a convenience sample based on review studies of Cagnie at al., 2015, and Espejo-Antúnez et al., 2017.

The study will be performed at the Laboratory of Evaluation and Rehabilitation of the Locomotor Apparatus (LARAL), located at Universidade Federal de Santa Catarina, Campus Araranguá, Santa Catarina, Brazil. Women, with age between 18 and 65 years old, students, workers, and professors at Universidade Federal de Santa Catarina (UFSC) will be invited to participate in the research. The invitation of subjects to participate in the study will be done through digital and printed folders that will be delivered at UFSC and on the social media. Those subjects that show interest to participate will be forwarded to an evaluation selection where it will be identified if the participant fits the inclusion criteria and where the Consent Form will be presented.

The active trigger point in upper trapezius will be localized through manual palpation and the location will be marked with a special pen for the skin. A second mark located 1.5 centimeters medially from the trigger point will be made in all subjects. The trigger point identification will follow Simons et al. criteria, featuring 3 of 4itens: (1) presence of palpable taut band in the muscle; (2) presence of hypersensitive spot inside the taut band; (3) subject recognize the familiar pain; and (4) painful limitation of the range of motion during total stretch.

The surface electromyography (EMG) will be used to evaluate the muscle recruitment pattern. Disposable electrodes, made with polyethylene foam and with hypoallergenic adhesive, solid gel adherent, bipolar contact of Silver/Silver Chloride (Ag/AgCl), will be used and positioned with 20mm of distance between poles. The Medtrace® reference electrode will be positioned in the ipsilateral wrist of the data collection. The electrodes will be positioned in the upper trapezius muscle as recommended by Surface ElectroMyoGraphy for the Non-Invasive Assessment of Muscles (SENIAM).

The Visual Analogue Scale (VAS) will be used so the subjects can graduate their pain in shoulder and neck regions. The VAS level of pain will be acquired before the intervention, soon after the intervention, 30 minutes after the intervention, one week and one month after the intervention.

Pressure algometry will be used to evaluate the pain pressure threshold (PPT). This measured will be obtained before the intervention (baseline), soon after the intervention, and 30 minutes after the intervention. The equipment will be positioned on the trigger point mark and the subject will be instructed to report when the sensation changes from pressure to pain. The force measured in kilograms per square centimeter (kg / cm²) will correspond to the quantity of pressure needed so the subject report change in pressure pain sensation.

The Neck Disability Index (NDI) is a unidimensional questionnaire composed of 10 items that have the aim to evaluate the limitation caused by pain and disability on the neck (30). This questionnaire will be self-applied and the subject will answer it before the intervention, one week and one month after intervention.

The Dry Needling (DN) protocol will be performed in one session. It will be used acupuncture needles, individually packaged and sterilized, with 0.25 mm of thickness and 0.40 mm of length. The therapist, then, will perform the grip in upper trapezius on the site of one of the two previously marked locations, according to the subject group allocation, and will insert the needle in the skin with help of a guide tube and will deepen the needle approximately 10 to 15 mm inside the trigger point. The needle will be moved up and down as in the "fast-in and fast-out" technique described by Hong. The movement will be repeated during 30 seconds in a cadence of approximately 1 Hz. The protocol will be the same for the groups that will receive the application directly on the trigger point and for the group that will receive the application away from the trigger point.

The photobiomodulation protocol will be performed using an equipment from Ibramed Equipamentos Médicos® of Aluminized Gallium Arsenide (AsGaAl) laser diode, with a wavelength of 830 nm, fluency of 20 J/cm², 30 milliwatts (mW), beam area of 0.116 cm², energy of 2,3 J per point, continuous beam. The low-level laser therapy (LLLT) will be applied for 30 seconds at one point on the trigger point in upper trapezius, right after the dry needling application.

The placebo/control group will receive the DN application 1.5 cm away from the trigger point and will follow the application protocol described above. The LLLT equipment will be turned off during the intervention. As the other groups, it will be performed one session of the dry needling followed by the intervention with the laser turned off.

The present study is grounded on the ethical principles, with base on the Resolution no 466 of December 12th, 2012, of the National Health Council, which incorporates under the individual and collectivities optics, the four basic references of the bioethics: autonomy, non-maleficence, beneficence, and justice, among others, aiming to ensure the rights and duties which concern the scientific community, the research subjects, and the State.

Data analysis will be performed through the GraphPad Prisma® software, version 6.01 (GraphPad Software, La Jolla, California, USA). The Shapiro-Wilk test will be run to verify sample normality distribution. The Two-Way ANOVA test will be used for comparative analysis inter and intra-groups. The P value (p<0.05) will be used to establish the significance of the results, in addition to the 95% Confidence Interval (95% CI). The values will be described as a mean ± standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* Presence of active trigger point in upper trapezius.
* Use of computer for typing activities for, at least, 20 hours per week.
* Presence of mechanic pain in cervical region for less than three months.
* Pain level higher than 3 and lower than 8 on the Visual Analogue Scale (VAS) for neck and cervical regions in the last 30 days.

Exclusion Criteria:

* Body Mass Index (BMI) higher than 30
* Presence of whiplash injury or other cervical pathologies such as herniated disc and
* Thoracic Gorge Syndrome;
* Presence of contraindication to the treatment with low-level laser therapy or with dry needling
* Fear of needles
* To be receiving treatment for the pain in neck and/or shoulder regions
* Make use of analgesic drugs, anti-inflammatory and/or muscle relaxants and anticoagulant medications.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Pain through the visual analogue scale at baseline | Measure will be obtained before the intervention (baseline).
  The Visual Analogue Scale (VAS) will be used so the subjects can graduate their pain in shoulder and neck regions. The scale range goes from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Pain through the visual analogue scale after 30 minutes of intervention | Measure will be obtained 30 minutes after the intervention
  The Visual Analogue Scale (VAS) will be used so the subjects can graduate their pain in shoulder and neck regions. The scale range goes from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Pain through the visual analogue scale after one week of intervention | Measure will be obtained 1 week after the intervention
  The Visual Analogue Scale (VAS) will be used so the subjects can graduate their pain in shoulder and neck regions. The scale range goes from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Pain through the visual analogue scale after one month of intervention | Measure will be obtained 30 days after the intervention
  The Visual Analogue Scale (VAS) will be used so the subjects can graduate their pain in shoulder and neck regions. The scale range goes from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.

SECONDARY OUTCOMES:
Pain Pressure Threshold | This measured will be obtained before the intervention (baseline)
  Measured through Pressure Algometry. The force measured in kilograms per square centimeter (kg / cm²) will correspond to the quantity of pressure needed so the subject report change in pressure pain sensation.
Pain Pressure Threshold | This measured will be obtained soon after the intervention (T1)
  Measured through Pressure Algometry. The force measured in kilograms per square centimeter (kg / cm²) will correspond to the quantity of pressure needed so the subject report change in pressure pain sensation.
Pain Pressure Threshold | This measured will be obtained 30 minutes after the intervention (T2)
  Measured through Pressure Algometry. The force measured in kilograms per square centimeter (kg / cm²) will correspond to the quantity of pressure needed so the subject report change in pressure pain sensation.
Muscle activity | Electromyographic data will be collected before the intervention and 5 minutes after the intervention.
  Electromyography will be used to measure muscle activity on upper trapezius
Functional Capacity | The subject will answer the NDI before the intervention
  Neck Disability Index (NDI) will be used to access the functional capacity. Its score ranges from 0 to 50, where 0 to 4 is considered total capacity, 5 to 14 is mild incapacity, 15 to 24 is moderate incapacity, 25 to 34 is serious incapacity, and >35 is severe incapacity.
Functional Capacity | The subject will answer the NDI 1 week after intervention
  Neck Disability Index (NDI) will be used to access the functional capacity. Its score ranges from 0 to 50, where 0 to 4 is considered total capacity, 5 to 14 is mild incapacity, 15 to 24 is moderate incapacity, 25 to 34 is serious incapacity, and >35 is severe incapacity.
Functional Capacity | The subject will answer the NDI 1 month after intervention
  Neck Disability Index (NDI) will be used to access the functional capacity. Its score ranges from 0 to 50, where 0 to 4 is considered total capacity, 5 to 14 is mild incapacity, 15 to 24 is moderate incapacity, 25 to 34 is serious incapacity, and >35 is severe incapacity.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael I Barbosa, PhD, Principal Investigator — Universidade Federal de Santa Catarina
Locations (1):
- Universidade Federal de Santa Catarina, Araranguá, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data that underlie results in a publication will be available after the end of the study for researchers that have doubts about it.
Supporting Information: Study Protocol
Time Frame: Study protocol will be submitted for publication before the end of the study.
Access Criteria: To be a principal researcher associated with a higher education institution.

REFERENCES:
- [Background] Boyles R, Fowler R, Ramsey D, Burrows E. Effectiveness of trigger point dry needling for multiple body regions: a systematic review. J Man Manip Ther. 2015 Dec;23(5):276-93. doi: 10.1179/2042618615Y.0000000014. PMID 26955257
- [Background] Kamanli A, Kaya A, Ardicoglu O, Ozgocmen S, Zengin FO, Bayik Y. Comparison of lidocaine injection, botulinum toxin injection, and dry needling to trigger points in myofascial pain syndrome. Rheumatol Int. 2005 Oct;25(8):604-11. doi: 10.1007/s00296-004-0485-6. Epub 2004 Sep 15. PMID 15372199
- [Background] Ge HY, Arendt-Nielsen L, Farina D, Madeleine P. Gender-specific differences in electromyographic changes and perceived pain induced by experimental muscle pain during sustained contractions of the upper trapezius muscle. Muscle Nerve. 2005 Dec;32(6):726-33. doi: 10.1002/mus.20410. PMID 16136601
- [Background] Mata Diz JB, de Souza JR, Leopoldino AA, Oliveira VC. Exercise, especially combined stretching and strengthening exercise, reduces myofascial pain: a systematic review. J Physiother. 2017 Jan;63(1):17-22. doi: 10.1016/j.jphys.2016.11.008. Epub 2016 Dec 3. PMID 27989732
- [Background] Dunning J, Butts R, Mourad F, Young I, Flannagan S, Perreault T. Dry needling: a literature review with implications for clinical practice guidelines. Phys Ther Rev. 2014 Aug;19(4):252-265. doi: 10.1179/108331913X13844245102034. PMID 25143704
- [Background] Espejo-Antunez L, Tejeda JF, Albornoz-Cabello M, Rodriguez-Mansilla J, de la Cruz-Torres B, Ribeiro F, Silva AG. Dry needling in the management of myofascial trigger points: A systematic review of randomized controlled trials. Complement Ther Med. 2017 Aug;33:46-57. doi: 10.1016/j.ctim.2017.06.003. Epub 2017 Jun 15. PMID 28735825
- [Background] Ilbuldu E, Cakmak A, Disci R, Aydin R. Comparison of laser, dry needling, and placebo laser treatments in myofascial pain syndrome. Photomed Laser Surg. 2004 Aug;22(4):306-11. doi: 10.1089/pho.2004.22.306. PMID 15345173
- [Background] Manca A, Limonta E, Pilurzi G, Ginatempo F, De Natale ER, Mercante B, Tolu E, Deriu F. Ultrasound and laser as stand-alone therapies for myofascial trigger points: a randomized, double-blind, placebo-controlled study. Physiother Res Int. 2014 Sep;19(3):166-75. doi: 10.1002/pri.1580. Epub 2014 Jan 2. PMID 24382836
- [Background] Hong CZ. Treatment of myofascial pain syndrome. Curr Pain Headache Rep. 2006 Oct;10(5):345-9. doi: 10.1007/s11916-006-0058-3. PMID 16945250
- [Background] Pecos-Martin D, Montanez-Aguilera FJ, Gallego-Izquierdo T, Urraca-Gesto A, Gomez-Conesa A, Romero-Franco N, Plaza-Manzano G. Effectiveness of dry needling on the lower trapezius in patients with mechanical neck pain: a randomized controlled trial. Arch Phys Med Rehabil. 2015 May;96(5):775-81. doi: 10.1016/j.apmr.2014.12.016. Epub 2015 Jan 9. PMID 25582412
- [Background] Uemoto L, Nascimento de Azevedo R, Almeida Alfaya T, Nunes Jardim Reis R, Depes de Gouvea CV, Cavalcanti Garcia MA. Myofascial trigger point therapy: laser therapy and dry needling. Curr Pain Headache Rep. 2013 Sep;17(9):357. doi: 10.1007/s11916-013-0357-4. PMID 23904202
- [Background] Cotler HB, Chow RT, Hamblin MR, Carroll J. The Use of Low Level Laser Therapy (LLLT) For Musculoskeletal Pain. MOJ Orthop Rheumatol. 2015;2(5):00068. doi: 10.15406/mojor.2015.02.00068. Epub 2015 Jun 9. PMID 26858986
- [Background] De Meulemeester K, Calders P, Dewitte V, Barbe T, Danneels L, Cagnie B. Surface Electromyographic Activity of the Upper Trapezius Before and After a Single Dry Needling Session in Female Office Workers With Trapezius Myalgia. Am J Phys Med Rehabil. 2017 Dec;96(12):861-868. doi: 10.1097/PHM.0000000000000761. PMID 28644247
- [Background] Mejuto-Vazquez MJ, Salom-Moreno J, Ortega-Santiago R, Truyols-Dominguez S, Fernandez-de-Las-Penas C. Short-term changes in neck pain, widespread pressure pain sensitivity, and cervical range of motion after the application of trigger point dry needling in patients with acute mechanical neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Apr;44(4):252-60. doi: 10.2519/jospt.2014.5108. Epub 2014 Feb 25. PMID 24568260

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT03375229/Prot_SAP_ICF_001.pdf